CLINICAL TRIAL: NCT04090073
Title: Electroacupuncture Combined With Fast-track Perioperative Program for Reducing Duration of Postoperative Ileus and Hospital Stay After Laparoscopic Colorectal Surgery: A Randomized Controlled Trial
Brief Title: Electroacupuncture Combined With Fast-track Perioperative Program for Laparoscopic Colorectal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon S. M. Ng, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CREC 2017.668-T
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture Plus Fast-track Perioperative Program (Experimental): Patients who are randomized to the intervention arm will receive Electroacupuncture combined with Fast-track program. Each session of Electroacupuncture will last for 20 minutes. The patients will undergo one session of Electroacupuncture daily from day 1 till day 4, or until the time when the primary outcome has occurred, whichever is earlier.
  Interventions: Procedure: Electroacupuncture; Other: Fast-track Perioperative program
- Fast-track Perioperative Program (Active Comparator): Patients who are randomized to the control arm will receive Fast-track program alone.
  Interventions: Other: Fast-track Perioperative program

INTERVENTIONS:
Procedure: Electroacupuncture — As above
  Arms: Electroacupuncture Plus Fast-track Perioperative Program
Other: Fast-track Perioperative program — As above

SUMMARY:
Background: The investigators' previous study demonstrated that electroacupuncture (EA) reduces the duration of postoperative ileus and hospital stay after laparoscopic colorectal surgery within a traditional perioperative care setting. Recent evidence also suggested that a 'fast-track' (FT) perioperative program may help accelerate recovery after colorectal surgery. It is uncertain whether the combination of EA and FT program will result in faster recovery after laparoscopic colorectal surgery when compared with FT program alone.

Objectives: To compare the efficacy of EA combined with FT program versus FT program alone in reducing the duration of postoperative ileus and hospital stay after laparoscopic colorectal surgery

Design: Prospective randomized trial.

Subjects: 72 consecutive patients undergoing elective laparoscopic resection of colonic and upper rectal cancer without conversion will be recruited.

Interventions: Patients will be randomly allocated to one of the two groups receiving either EA + FT program, or FT program alone.

Outcome measures: Primary outcome: time to defecation. Secondary outcomes: duration of hospital stay, time to resume diet, pain scores, analgesic requirement, morbidity, quality of life, and medical costs.

Conclusions: This study serves as a good example that illustrates an integrated approach in combining Chinese and Western models of health care. It will provide evidence-based clarification of the role of EA in enhancing recovery after laparoscopic colorectal surgery within a FT perioperative care setting. As laparoscopic colorectal surgery has been shown to have a higher direct cost than the open counterpart, a faster postoperative recovery may help reduce the financial burden to the hospital/healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing elective laparoscopic resection of colonic and upper rectal cancer (adenocarcinoma of the colorectum of which the lowest margin of the tumor is located >12 cm from the anal verge as measured by rigid sigmoidoscopy)
* Age of patients >18 years
* Those with American Society of Anesthesiologists (ASA) grading I-III
* Those with no cognitive impairment (Mini Mental State Examination score 24 out of 30)
* Those with no severe physical disability
* Those who require no assistance with the activities of daily living
* Informed consent available

Exclusion Criteria:

* Patients undergoing laparoscopic low anterior resection with total mesorectal excision, abdominoperineal resection, or total/proctocolectomy; those with planned stoma creation
* Those undergoing simultaneous laparoscopic resection of colorectal cancer and other coexisting intraabdominal diseases
* Those undergoing laparoscopic resection of colorectal cancer with en bloc resection of surrounding organs
* Those who developed intraoperative problems or complications that required conversion
* Those undergoing emergency surgery
* Those with evidence of peritoneal carcinomatosis
* Those with previous history of midline laparotomy
* Those who are expected to receive epidural opioids for postoperative pain management
* Those who are pregnant
* Those with cardiac pacemaker
* Those with coagulopathy
* Those who are allergic to the acupuncture needles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Time to defecation | Up to 1 month
  Measured in hours, from the time the laparoscopic surgery ends till the first observed passage of stool.

SECONDARY OUTCOMES:
Total postoperative hospital stay | Up to 1 month
  Including hospital stay of patients who are readmitted within 30 days after surgery
Time of first passing flatus reported by the patients | Up to 1 month
Time that the patients tolerated solid diet | Up to 1 month
  Time that the patients tolerated solid diet (any food that required chewing) without vomiting or experiencing significant nausea 4 hours following the meal
Time to walk independently | Up to 1 month
Pain scores on visual analog scale | Up to 1 month
  From 0 which implies no pain at all, to 100 which implies the worst pain imaginable, on the first 3 postoperative days
Postoperative 30-day morbidity | Up to 1 month
  Defined by the Clavien-Dindo classification of surgical complications
Incidence rate of adverse events related to electroacupuncture | Up to 1 month
Readmission rate | Up to 1 month
Quality of life scores measured by Short Form 36 (SF-36) Health Survey at 2 and 4 weeks after surgery | Up to 1 month
  SF-36 Health Survey is a 36-item, patient-reported survey of patient health. It consists of eight scaled scores, which are the weighted sums of the questions in their section. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of life scores measured by European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaires at 2 and 4 weeks after surgery | Up to 1 month
  EORTC QLQ-C30 is a generic questionnaire for assessment of quality of life (QoL) in cancer patients. It includes 30 items, 24 of which are combined to form a global QoL scale, five functional scales (physical, role, emotional, cognitive, and social), and three symptom scales (fatigue, nausea/vomiting, and pain). The other six single items evaluate dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties. All questionnaires responses and scores will be linearly transformed to a 0-100 scale. A higher score on the global QoL and functional scales represents a higher level of QoL and functioning, whereas a higher score on the symptom scales/items represents a higher degree of symptoms or dysfunction.
Quality of life measured by European Organisation for Research and Treatment of Cancer (EORTC) QLQ-CR38 questionnaires at 2 and 4 weeks after surgery | Up to 1 month
  EORTC QLQ-CR38 is a specific questionnaire module specifically designed for assessment of quality of life (QoL) in patients with colorectal cancer. It consists of 38 items covering symptoms and side effects related to different colorectal cancer treatment modalities. The module contains four functional scales (body image, sexual functioning, sexual enjoyment, and future perspective) and eight symptom scales/items (micturition problems, chemotherapy side effects, gastrointestinal tract symptoms, male sexual problems, female sexual problems, defecation problems, stoma-related problems, and weight loss). All questionnaires responses and scores will be linearly transformed to a 0-100 scale. A higher score on the global QoL and functional scales represents a higher level of QoL and functioning, whereas a higher score on the symptom scales/items represents a higher degree of symptoms or dysfunction.
Direct/indirect medical costs and out-of-hospital economic costs | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Simon SM Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No